CLINICAL TRIAL: NCT01265784
Title: A Phase 2, Randomized, Double-Blind, Double-Dummy, Multicenter, Prospective Study to Assess the Efficacy, Safety, and PK of 2 Dose Regimens of TP-434 Compared With Ertapenem in Adult Community-Acquired Complicated Intra-abdominal Infections
Brief Title: Study to Compare TP-434 and Ertapenem in Community-acquired Complicated Intra-abdominal Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-434-P2-cIAI-1
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Complicated Intra-abdominal Infection
MeSH Terms: interventions — eravacycline; Ertapenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TP-434, 1.5 mg/kg q24h (Experimental): TP-434 was administered intravenously (IV) at a dose of 1.5 milligrams per kilogram of body weight (mg/kg) every 24 hours (q24h) for a minimum of 4 days and a maximum of 14 days (7 days for participants in India). TP-434 treatment was to be stopped when symptoms of complicated intra-abdominal infection (cIAI) resolved, there was treatment failure, or the maximum allowed number of infusion days was reached.
  Interventions: Drug: TP-434; Drug: Placebo
- TP-434, 1.0 mg/kg q12h (Experimental): TP-434 was administered IV at a dose of 1.0 mg/kg every 12 hours (q12h) for a minimum of 4 days and a maximum of 14 days (7 days for participants in India). TP-434 treatment was to be stopped when symptoms of cIAI resolved, there was treatment failure, or the maximum allowed number of infusion days was reached.
  Interventions: Drug: TP-434; Drug: Placebo
- Ertapenem, 1 g q24h (Active Comparator): Ertapenem was administered IV at a dose of 1 gram (g) q24h for a minimum of 4 days and a maximum of 14 days (7 days for participants in India). Ertapenem treatment was to be stopped when symptoms of cIAI resolved, there was treatment failure, or the maximum allowed number of infusion days was reached.
  Interventions: Drug: Ertapenem; Drug: Placebo

INTERVENTIONS:
Drug: TP-434
  Other Names: Eravacycline
  Arms: TP-434, 1.0 mg/kg q12h; TP-434, 1.5 mg/kg q24h
Drug: Ertapenem
  Other Names: Invanz
  Arms: Ertapenem, 1 g q24h
Drug: Placebo — Administered IV to maintain the blind.

SUMMARY:
This is a Phase 2, randomized, double-blind, double-dummy, multicenter, prospective study to assess the efficacy, safety, and pharmacokinetics of two dose regimens of TP-434 compared with ertapenem in the treatment of adult community-acquired complicated intra-abdominal infections (cIAIs).

ELIGIBILITY:
Inclusion Criteria:

* Abdominal pain/discomfort with onset prior to hospitalization
* Evidence of a systemic inflammatory response
* Physical findings consistent with intra-abdominal infection (IAI)
* Clinical diagnosis of community-acquired IAI requiring urgent surgical or percutaneous intervention and not expected to require antibacterial therapy for longer than 14 days
* Body mass index (BMI) of ≤ 30 kilograms per square meter (kg/m^2)
* Able to provide informed consent. If the participant is unable to provide informed consent, the participant's legally acceptable representative may provide written consent in accordance with institutional guidelines
* If female, not pregnant or nursing or, if of child-bearing potential either: will commit to use at least two medically accepted, effective methods of birth control (for example, condom, oral contraceptive, indwelling intrauterine device, hormonal implant/patch, injections, approved cervical ring) during study drug dosing and for 90 days following last study drug dose or practicing sexual abstinence

Exclusion Criteria:

* Symptoms related to diagnosis of complicated appendicitis (if current diagnosis) for < 24 hours prior to current hospitalization
* Previously hospitalized or admitted to a healthcare facility within the last 6 months
* Managed by Staged Abdominal Repair or other open abdomen technique
* Known at study entry to have an IAI caused by a pathogen(s) resistant to both study drug antibiotics
* Acute Physiology and Chronic Health Evaluation (APACHE) II score > 25
* Unlikely to survive the 6-8 week study period
* Any rapidly-progressing disease or immediately life-threatening illness, including acute hepatic failure, respiratory failure and septic shock
* Requirement for vasopressors at therapeutic dosages
* Renal failure
* Presence or possible signs of hepatic disease
* Hematocrit < 25% or hemoglobin < 8 grams per deciliter (g/dL)
* Neutropenia with absolute neutrophil count < 1000 cells per cubic millimeter (mm^3)
* Platelet count < 50,000/mm3
* Abnormal coagulation tests or participant on anticoagulants
* Immunocompromised condition, including known human immunodeficiency virus (HIV) positivity or acquired immune deficiency syndrome (AIDS), organ (bone marrow) transplant recipients, and hematological malignancy. Immunosuppressive therapy, including use of high-dose corticosteroids (for example, > 40 milligrams [mg] prednisone or equivalent per day for greater than 2 weeks)
* History of hypersensitivity reactions to tetracyclines or carbapenems
* Participation in any investigational drug or device study within 30 days prior to study entry
* Known or suspected central nervous system (CNS) disorder that may predispose to seizures or lower seizure threshold
* Previously received TP-434 in a clinical trial
* More than 24 hours duration of systemic antibiotic coverage for current condition
* Received ertapenem or any other carbapenem, or tigecycline for the current infection
* Need for concomitant systemic antimicrobial agents other than study drug or received systemic (IV or oral) antibiotics in the last 3 months
* Refusal of mechanical ventilation, dialysis or hemofiltration, cardioversion or any other resuscitative measures and drug/fluid therapy at time of consent
* Known or suspected inflammatory bowel disease or associated visceral abscess

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Horn, MD, PhD, Study Director — Tetraphase Pharmaceuticals, Inc
Locations (38):
- United States (5):
  - Long Beach VA Medical Center, Long Beach, California
  - Denver Health Medical Center, Denver, Colorado
  - Henry Ford Hospital, Detroit, Michigan
  - Barnes Jewish Hospital, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
- Bulgaria (8):
  - MHAT "Yulia Vrevska - Byala" EOOD, Byala, Byala
  - UMHAT "Dr. Georgi Stranski" EAD, Pleven, Pleven
  - UMHAT "Sveti Georgi" EAD, Plovdiv, Plovdiv
  - MHAT "Russe" AD, Russe, Rousse
  - MHAT "Tokuda Hospital Sofia" AD, Sofia, Sofia
  - UMHAT "Tzaritza Yoanna" EAD, Sofia, Sofia
  - UMHATEM "N.I. Pirogov" EAD, Sofia, Sofia
  - UMHATEM "N.I.Pirogov" EAD, Sofia, Sofia
- India (9):
  - Bangalore Medical College and Research Institute, Victoria Hospital, Fort Mumbai, Bangalore
  - Amrita Institute of Medical Sciences and Research Centre, Kochi, Kerala
  - Sahyadri Munot Hospital, Pune, Maharashtra
  - S.R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - HCG-Medisurge Hospitals Pvt. Ltd., Ahmedabad
  - Santosh Hospital, Bangalore
  - K.R. Hospital, Bangalore
  - M.S. Ramalah Medical College and Hospitals, Bangalore
  - Sai Vani Hospitals, Ltd., Hyderabad
- Latvia (4):
  - Daugavpils Regional Hospital, Daugavpils
  - Jekabpils Regional Hospital, Jēkabpils
  - Rezeknes Hospital, Rēzekne
  - Vidzeme Hospital, Valmiera
- Lithuania (6):
  - Kaunas Hospital, Kaunas
  - Kaunas Clinical Hospital, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Vilnius University Hospital Santariskiu Clinics, Vilnius
  - Vilnius City Clinical Hospital, Vilnius
- Romania (6):
  - Emergency Clinical City Hospital, Timișoara, Timiș County
  - "Dr. Carol Davila" Clinical Nephrology Hospital General Surgery Clinic, Bucharest
  - Emergency Clinical Hospital Bucharest, Bucharest
  - Coltea Clinical Hospital, Bucharest
  - :Sfantul loan" Clinical Emergency Hospital, Bucharest
  - University Emergency Hospital Bucharest, Bucharest

REFERENCES:
- [Derived] Solomkin JS, Ramesh MK, Cesnauskas G, Novikovs N, Stefanova P, Sutcliffe JA, Walpole SM, Horn PT. Phase 2, randomized, double-blind study of the efficacy and safety of two dose regimens of eravacycline versus ertapenem for adult community-acquired complicated intra-abdominal infections. Antimicrob Agents Chemother. 2014;58(4):1847-54. doi: 10.1128/AAC.01614-13. Epub 2013 Dec 16. PMID 24342651

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was stratified by site of infection (complicated appendicitis versus all other diagnoses).
Groups:
- TP-434, 1.5 mg/kg q24h: TP-434 was administered intravenously (IV) at a dose of 1.5 milligrams per kilogram of body weight (mg/kg) every 24 hours (q24h) for a minimum of 4 days and a maximum of 14 days (7 days for participants in India).
- TP-434, 1.0 mg/kg q12h: TP-434 was administered IV at a dose of 1.0 mg/kg every 12 hours (q12h) for a minimum of 4 days and a maximum of 14 days (7 days for participants in India).
- Ertapenem, 1 g q24h: Ertapenem was administered IV at a dose of 1 gram (g) q24h for a minimum of 4 days and a maximum of 14 days (7 days for participants in India).
Period: Overall Study
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem, 1 g q24h
Started | 56 | 57 | 30
Received at Least 1 Dose of Study Drug | 54 (1 participant randomized to TP-434 1.5 mg/kg took ertapenem. Results are included in ertapenem arm.) | 56 | 29
Completed | 44 | 49 | 26
Not Completed | 12 | 8 | 4
Not completed — Lost to Follow-up | 5 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 5 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 3 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Incorrectly Randomized | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- TP-434, 1.5 mg/kg q24h: TP-434 was administered IV at a dose of 1.5 mg/kg q24h for a minimum of 4 days and a maximum of 14 days (7 days for participants in India).
- TP-434, 1.0 mg/kg q12h: TP-434 was administered IV at a dose of 1.0 mg/kg q12h for a minimum of 4 days and a maximum of 14 days (7 days for participants in India).
- Ertapenem 1 g q24h: Ertapenem was administered IV at a dose of 1 g q24h for a minimum of 4 days and a maximum of 14 days (7 days for participants in India).
- Total: Total of all reporting groups
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h | Total
Number analyzed (Participants) | 56 | 57 | 30 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (18.39) | 42.1 (17.16) | 41.8 (17.60) | 42.6 (17.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 8 | 40
  Male | 38 | 43 | 22 | 103
Region of Enrollment [Number; unit: participants]
  United States | 0 | 0 | 1 | 1
  Romania | 6 | 9 | 6 | 21
  Lithuania | 17 | 13 | 7 | 37
  Bulgaria | 9 | 6 | 3 | 18
  Latvia | 8 | 9 | 4 | 21
  India | 16 | 20 | 9 | 45

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to TP-434 and Ertapenem in the Microbiologically Evaluable (ME) Population at the Test-of-Cure Visit
Description: Clinical response was classified as cure (complete resolution or significant improvement of signs and symptoms of the index infection), failure (death related to complicated intra-abdominal infection [cIAI], persisting or recurrent infection within the abdomen, postsurgical wound infection, or administration of effective concomitant antibacterial therapy), or indeterminate (Test-of-Cure [TOC] assessment was not available, death unrelated to cIAI, or some other reason).
Time Frame: TOC Visit (10-14 days after last dose of study drug)
Population: All randomized participants who received at least 1 dose of study drug, met the minimal disease definition of cIAI, had a baseline pathogen identified, and had a microbiological response assessed.
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 42 | 41 | 26
participants
  Cure | 39 | 41 | 24
  Failure | 3 | 0 | 2
  Indeterminate | 0 | 0 | 0

2. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Modified Intent-to-treat (MITT) Population at the End-of-Treatment (EOT) Visit
Time Frame: EOT Visit (4-14 days after first dose of study drug)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 54 | 56 | 29
participants
  Cure | 49 | 52 | 28
  Failure | 2 | 1 | 1
  Indeterminate | 3 | 3 | 0

3. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Modified Intent-to-treat (MITT) Population at TOC Visit
Time Frame: TOC Visit (10-14 days after last dose of study drug)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 54 | 56 | 29
participants
  Cure | 46 | 47 | 26
  Failure | 3 | 1 | 2
  Indeterminate | 5 | 8 | 1

4. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Modified Intent-to-treat (MITT) Population at the Follow-up Visit
Time Frame: Follow-up Visit (28-42 days after last dose of study drug)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 54 | 56 | 29
participants
  Cure | 41 | 45 | 24
  Failure | 4 | 1 | 2
  Indeterminate | 9 | 10 | 3

5. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Clinically Modified Intent-to-treat (c-MITT) Population at the EOT Visit
Time Frame: EOT Visit (4-14 days after first dose of study drug)
Population: All randomized participants who received at least 1 dose of study drug and met the minimal disease definition of intra-abdominal infection (IAI). The minimal disease definition included all IAI, whether complicated or not. Identification of a baseline pathogen was not required for this population.
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 54 | 56 | 29
participants
  Cure | 49 | 52 | 28
  Failure | 2 | 1 | 1
  Indeterminate | 3 | 3 | 0

6. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Clinically Modified Intent-to-treat (c-MITT) Population at the TOC Visit
Time Frame: TOC Visit (10-14 days after last dose of study drug)
Population: All randomized participants who received at least 1 dose of study drug and met the minimal disease definition of IAI. The minimal disease definition included all IAI, whether complicated or not. Identification of a baseline pathogen was not required for this population.
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 54 | 56 | 29
participants
  Cure | 46 | 47 | 26
  Failure | 3 | 1 | 2
  Indeterminate | 5 | 8 | 1

7. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Clinically Modified Intent-to-treat (c-MITT) Population at the Follow-up Visit
Time Frame: Follow-up Visit (28-42 days after last dose of study drug)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 54 | 56 | 29
participants
  Cure | 41 | 45 | 24
  Failure | 4 | 1 | 2
  Indeterminate | 9 | 10 | 3

8. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Microbiologically Modified Intent-to-treat (m-MITT) Population at the EOT Visit
Time Frame: EOT Visit (4-14 days after first dose of study drug)
Population: All randomized participants who received at least 1 dose of study drug, met the minimal disease definition of cIAI, and had a baseline pathogen identified. The minimal disease definition of cIAI included IAI that extended beyond the hollow viscus of origin into the peritoneal space and was associated with either abscess formation or peritonitis.
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 45 | 47 | 27
participants
  Cure | 41 | 44 | 26
  Failure | 2 | 0 | 1
  Indeterminate | 2 | 3 | 0

9. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Microbiologically Modified Intent-to-treat (m-MITT) Population at the TOC Visit
Time Frame: TOC Visit (10-14 days after last dose of study drug)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 45 | 47 | 27
participants
  Cure | 39 | 41 | 24
  Failure | 3 | 0 | 2
  Indeterminate | 3 | 6 | 1

10. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Microbiologically Modified Intent-to-treat (m-MITT) Population at the Follow-up Visit
Time Frame: Follow-Up Visit (28-42 days after last dose of study drug)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 45 | 47 | 27
participants
  Cure | 36 | 39 | 22
  Failure | 4 | 0 | 2
  Indeterminate | 5 | 8 | 3

11. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Clinically Evaluable (CE) Population at the EOT Visit
Time Frame: EOT Visit (4-14 days after first dose of study drug)
Population: All randomized participants who received at least 1 dose of study drug, met the minimal disease definition of cIAI, and for whom sufficient information was available to determine the participant's outcome with no confounding factors present that interfered with the assessment of that outcome.
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 49 | 48 | 28
participants
  Cure | 47 | 47 | 27
  Failure | 2 | 1 | 1
  Indeterminate | 0 | 0 | 0

12. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Clinically Evaluable (CE) Population at the TOC Visit
Time Frame: TOC Visit (10-14 days after last dose of study drug)
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 49 | 48 | 28
participants
  Cure | 46 | 47 | 26
  Failure | 3 | 1 | 2
  Indeterminate | 0 | 0 | 0

13. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Clinically Evaluable (CE) Population at the Follow-up Visit
Time Frame: Follow-up Visit (28-42 days after last dose of study drug)
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 49 | 48 | 28
participants
  Cure | 41 | 45 | 23
  Failure | 4 | 1 | 2
  Indeterminate | 4 | 2 | 3

14. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Microbiologically Evaluable (ME) Population at the EOT Visit
Time Frame: EOT Visit (4-14 days after first dose of study drug)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 42 | 41 | 26
participants
  Cure | 40 | 41 | 25
  Failure | 2 | 0 | 1
  Indeterminate | 0 | 0 | 0

15. Secondary Outcome: Clinical Response to TP-434 and Ertapenem in the Microbiologically Evaluable (ME) Population at the Follow-up Visit
Time Frame: Follow-up Visit (28-42 days after last dose of study drug)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 42 | 41 | 26
participants
  Cure | 36 | 39 | 21
  Failure | 4 | 0 | 2
  Indeterminate | 2 | 2 | 3

16. Secondary Outcome: Microbiologic Response to TP-434 and Ertapenem in the m-MITT Population at the EOT Visit
Description: Microbiological response was classified as favorable (eradication or presumed eradication), unfavorable (persistence, presumed persistence, superinfection, or new infection), or indeterminate (assessment not possible).
Time Frame: EOT Visit (4-14 days after first dose of study drug)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 45 | 47 | 27
participants
  Favorable | 41 | 44 | 26
  Unfavorable | 2 | 0 | 1
  Indeterminate | 2 | 3 | 0

17. Secondary Outcome: Microbiologic Response to TP-434 and Ertapenem in the m-MITT Population at the TOC Visit
Time Frame: TOC Visit (10-14 days after last dose of study drug)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 45 | 47 | 27
participants
  Favorable | 39 | 42 | 24
  Unfavorable | 3 | 0 | 2
  Indeterminate | 3 | 5 | 1

18. Secondary Outcome: Microbiologic Response to TP-434 and Ertapenem in the ME Population at the EOT Visit
Time Frame: EOT Visit (4-14 days after first dose of study drug)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 42 | 41 | 26
participants
  Favorable | 40 | 41 | 25
  Unfavorable | 2 | 0 | 1
  Indeterminate | 0 | 0 | 0

19. Secondary Outcome: Microbiologic Response to TP-434 and Ertapenem in the ME Population at the TOC Visit
Time Frame: TOC Visit (10-14 days after last dose of study drug)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Number analyzed (Participants) | 42 | 41 | 26
participants
  Favorable | 39 | 41 | 24
  Unfavorable | 3 | 0 | 2
  Indeterminate | 0 | 0 | 0

20. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of TP-434
Time Frame: Prior to first infusion and 1, 3, 7, 12, 48, and 108 hours after start of first infusion
Population: All randomized participants without significant protocol deviations who received at least 1 dose of TP-434 and had evaluable Cmax data.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h
Number analyzed (Participants) | 48 | 51
nanograms per milliliter (ng/mL) | 1445.625 (1168.029) | 952.608 (759.754)

21. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve From Time 0 to 12 Hours (AUC[0-12]) of TP-434
Time Frame: Prior to first infusion and 1, 3, 7, 12, 48, and 108 hours after start of first infusion
Population: All randomized participants without significant protocol deviations who received at least 1 dose of TP-434 and had evaluable AUC(0-12) data.
Measure: Mean (Standard Deviation); unit: nanogram*hours per milliliter (ng*h/mL)
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h
Number analyzed (Participants) | 48 | 47
nanogram*hours per milliliter (ng*h/mL) | 4349.900 (2186.791) | 3240.724 (1732.172)

ADVERSE EVENTS:
Arm/Group | TP-434, 1.5 mg/kg q24h | TP-434, 1.0 mg/kg q12h | Ertapenem 1 g q24h
Serious Adverse Events (participants affected / at risk) | 6/53 | 1/56 | 1/30
Other Adverse Events (participants affected / at risk) | 11/53 | 10/56 | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TP-434, 1.5 mg/kg q24h (N=53) | TP-434, 1.0 mg/kg q12h (N=56) | Ertapenem 1 g q24h (N=30)
Lobar Pneumonia (Infections and infestations) | 1 | 0 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 — Resulted in 1 death
Abdominal Wall Abscess (Infections and infestations) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 — Resulted in 1 death
Embolism (Vascular disorders) | 1 | 0 | 0 — Resulted in 1 death
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 1 | 0
Subdiaphragmatic Abscess (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TP-434, 1.5 mg/kg q24h (N=53) | TP-434, 1.0 mg/kg q12h (N=56) | Ertapenem 1 g q24h (N=30)
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 6 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0
Application Site Hypersensitivity (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Blood Amylase Increased (Investigations) | 3 | 2 | 1
Lipase Increased (Investigations) | 3 | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days prior to submitting or presenting a manuscript, poster, presentation, abstract or other materials relating to the Trial, the PI shall provide to Sponsor all such manuscripts and materials, and Sponsor shall have 60 days to review and comment. If requested, the PI shall remove Confidential lnformation prior to submitting or presenting the materials, and shall delay publication or presentation for up to 90 days to allow Sponsor to protect its interests in any such materials.